CLINICAL TRIAL: NCT02754765
Title: Evaluating Newly Approved Drugs for Multidrug-resistant TB (endTB): A Clinical Trial
Brief Title: Evaluating Newly Approved Drugs for Multidrug-resistant TB
Acronym: endTB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Médecins Sans Frontières, France (Other)
Collaborators: Partners in Health (Other); Harvard Medical School (HMS and HSDM) (Other); Epicentre (Other); Institute of Tropical Medicine, Belgium (Other); Socios En Salud, Peru (Unknown); Interactive Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSF ERB-1555
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Tuberculosis, Multidrug-Resistant; Infection, Bacterial; Pulmonary Tuberculoses
Keywords: bedaquiline; delamanid; linezolid; clofazimine; tuberculosis; MDR-TB XDR-TB
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Bacterial Infections; Tuberculosis, Pulmonary; Tuberculosis | interventions — bedaquiline; OPC-67683; Clofazimine; Levofloxacin; Moxifloxacin; Linezolid; Pyrazinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- endTB regimen 1 (BeLiMoZ) (Experimental): Subjects who are randomized to this arm will receive treatment for 39 weeks and post-treatment followup for 65 weeks. Participants may take as long as 47 weeks to complete all doses of a 39-week treatment regimen. Dosing of experimental regimens will be oral and weight based. Subjects will undergo a linezoilid dose reduction randomization to either 300mg daily or 600mg three times a week after 16 weeks of treatment or after a linezolid-related AE requiring dose reduction, whichever is earlier.
  Interventions: Drug: Bedaquiline; Drug: Moxifloxacin; Drug: Linezolid; Drug: Pyrazinamide
- endTB regimen 2 (BeLiCLeZ) (Experimental): Subjects who are randomized to this arm will receive treatment for 39 weeks and post-treatment followup for 65 weeks. Participants may take as long as 47 weeks to complete all doses of a 39-week treatment regimen. Dosing of experimental regimens will be oral and weight based. Subjects will undergo a linezoilid dose reduction randomization to either 300mg daily or 600mg three times a week after 16 weeks of treatment or after a linezolid-related AE requiring dose reduction, whichever is earlier.
  Interventions: Drug: Bedaquiline; Drug: Clofazimine; Drug: Levofloxacin; Drug: Linezolid; Drug: Pyrazinamide
- endTB regimen 3 (BeDeLiLeZ) (Experimental): Subjects who are randomized to this arm will receive treatment for 39 weeks and post-treatment followup for 65 weeks. Participants may take as long as 47 weeks to complete all doses of a 39-week treatment regimen. Dosing of experimental regimens will be oral and weight based. Subjects will undergo a linezoilid dose reduction randomization to either 300mg daily or 600mg three times a week after 16 weeks of treatment or after a linezolid-related AE requiring dose reduction, whichever is earlier.
  Interventions: Drug: Bedaquiline; Drug: Delamanid; Drug: Levofloxacin; Drug: Linezolid; Drug: Pyrazinamide
- endTB regimen 4 (DeLiCLeZ) (Experimental): Subjects who are randomized to this arm will receive treatment for 39 weeks and post-treatment followup for 65 weeks. Participants may take as long as 47 weeks to complete all doses of a 39-week treatment regimen. Dosing of experimental regimens will be oral and weight based. Subjects will undergo a linezoilid dose reduction randomization to either 300mg daily or 600mg three times a week after 16 weeks of treatment or after a linezolid-related AE requiring dose reduction, whichever is earlier.
  Interventions: Drug: Delamanid; Drug: Clofazimine; Drug: Levofloxacin; Drug: Linezolid; Drug: Pyrazinamide
- endTB regimen 5 (DeCMoZ) (Experimental): Subjects who are randomized to this arm will receive treatment for 39 weeks and post-treatment followup for 65 weeks. Participants may take as long as 47 weeks to complete all doses of a 39-week treatment regimen. Dosing of experimental regimens will be oral and weight based.
  Interventions: Drug: Delamanid; Drug: Clofazimine; Drug: Moxifloxacin; Drug: Pyrazinamide
- endTB regimen 6 (Control) (Active Comparator): endTB regimen 6 is the control regimen.
  Interventions: Drug: Control arm MDR-TB regimen, consistent with WHO guidelines

INTERVENTIONS:
Drug: Bedaquiline
  Other Names: Sirturo
  Arms: endTB regimen 1 (BeLiMoZ); endTB regimen 2 (BeLiCLeZ); endTB regimen 3 (BeDeLiLeZ)
Drug: Delamanid
  Other Names: Deltyba; OPC-67683
  Arms: endTB regimen 3 (BeDeLiLeZ); endTB regimen 4 (DeLiCLeZ); endTB regimen 5 (DeCMoZ)
Drug: Clofazimine
  Other Names: Lamprene
  Arms: endTB regimen 2 (BeLiCLeZ); endTB regimen 4 (DeLiCLeZ); endTB regimen 5 (DeCMoZ)
Drug: Levofloxacin
  Arms: endTB regimen 2 (BeLiCLeZ); endTB regimen 3 (BeDeLiLeZ); endTB regimen 4 (DeLiCLeZ)
Drug: Moxifloxacin
  Arms: endTB regimen 1 (BeLiMoZ); endTB regimen 5 (DeCMoZ)
Drug: Linezolid
  Arms: endTB regimen 1 (BeLiMoZ); endTB regimen 2 (BeLiCLeZ); endTB regimen 3 (BeDeLiLeZ); endTB regimen 4 (DeLiCLeZ)
Drug: Pyrazinamide
  Arms: endTB regimen 1 (BeLiMoZ); endTB regimen 2 (BeLiCLeZ); endTB regimen 3 (BeDeLiLeZ); endTB regimen 4 (DeLiCLeZ); endTB regimen 5 (DeCMoZ)
Drug: Control arm MDR-TB regimen, consistent with WHO guidelines — Control arm MDR-TB regimen, consistent WHO guidelines
  Arms: endTB regimen 6 (Control)

SUMMARY:
endTB Clinical Trial a Phase III, randomized, controlled, open-label, non-inferiority, multi-country trial evaluating the efficacy and safety of five new, all-oral, shortened regimens for multidrug-resistant tuberculosis (MDR-TB).

DETAILED DESCRIPTION:
This is a Phase III, randomized, controlled, open-label, non-inferiority, multi-country trial evaluating the efficacy and safety of new combination regimens for MDR-TB treatment.

Regimens examined combine newly approved drugs bedaquiline and/or delamanid with existing drugs known to be active against Mycobacterium tuberculosis (linezolid, clofazimine, moxifloxacin or levofloxacin, and pyrazinamide). The study will enroll in parallel across 5 experimental and 1 standard-of-care control arms. Randomization will be outcome adapted using Bayesian interim analysis of efficacy endpoints. Experimental regimens will contain bedaquiline and/or delamanid and up to 4 companion drugs. Control-arm treatment may contain one of the following (bedaquiline or delamanid) and companion drugs, constructed and delivered according to local standard of care and consistent with WHO guidelines. Trial participation in all arms will last at least until Week 73, and up to Week 104. In the experimental arms, treatment will be for 39 weeks (participants in the experimental arms will be allowed up to 47 weeks to complete the 39-week treatment course) and post-treatment follow up for up to 65 additional weeks. In the control arm, treatment will be delivered according to local standard of care (in consistence with WHO guidance); duration may vary and will be approximately 86 weeks for the conventional regimen and 39-52 weeks for the standardized shorter regimen.

Non-inferiority will be established for any experimental arm if the lower bound of the one-sided 97.5% confidence interval around the difference in favorable outcome between the control and experimental arms is greater than or equal to -12%.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for randomization if s/he:

1. Has documented pulmonary tuberculosis due to strains of M. tuberculosis resistant to rifampin (RIF) and susceptible to fluoroquinolones, diagnosed by validated rapid molecular test;
2. Is ≥ 15 years of age;
3. Is willing to use contraception: pre-menopausal women or women whose last menstrual period was within the preceding year, who have not been sterilized must agree to use contraception unless their partner has had a vasectomy; men who have not had a vasectomy must agree to use condoms;
4. Provides informed consent for study participation; additionally a legal representative of patients considered minor per local laws should also provide consent;
5. Lives in a dwelling that can be located by study staff and expects to remain in the area for the duration of the study.

Exclusion Criteria:

A patient will not be eligible for randomization if s/he:

1. Has known allergies or hypersensitivity to any of the investigational drugs;
2. Is known to be pregnant or is unwilling or unable to stop breast-feeding an infant;
3. Is unable to comply with treatment or follow-up schedule;
4. Any condition (social or medical) which, in the opinion of the site principal investigator, would make study participant unsafe;
5. a. Has had exposure (intake of the drug for 30 days or more) in the past five years to bedaquiline, delamanid, linezolid, or clofazimine, or has proven or likely resistance to bedaquiline, delamanid, linezolid, or clofazimine (e.g., household contact of a DR-TB index case who died or experienced treatment failure after treatment containing bedaquiline, delamanid, linezolid, or clofazimine or had resistance to one of the listed drugs); exposure to other anti-TB drugs is not a reason for exclusion.

   b. Has received second-line drugs for 15 days or more prior to screening visit date in the current MDR/RR-TB treatment episode. Exceptions include: (1) patients whose treatment has failed according to the WHO definition151 and who are being considered for a new treatment regimen; (2) patients starting a new treatment regimen after having been "lost to follow-up" according to the WHO definition149 and, (3) patients in whom treatment failure is suspected (but not confirmed according to WHO definition), who are being considered for a new treatment regimen, and for whom the Clinical Advisory Committee (CAC) consultation establishes eligibility.
6. Has one or more of the following:

   * Hemoglobin ≤ 7.9 g/dL;
   * Uncorrectable electrolytes disorders:
   * Calcium < 7.0 mg/dL;
   * Potassium < 3.0 or ≥6.0 mEq/L;
   * Magnesium < 0.9 mEq/L;
   * Serum creatinine > 3 x ULN;
   * Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) ≥ 3 x ULN;
   * Total bilirubin ≥ 1.5 x ULN if accompanied by AST or ALT > ULN or total bilirubin ≥ 2 x ULN when other liver function results are in the normal range;
   * Grade 4 result on any of the specified laboratory tests as defined by the MSF Severity Scale.
7. Has cardiac risk factors defined as:

   * A confirmed QTc interval of greater than or equal to 450 ms. Retesting to reassess eligibility will be allowed once using an unscheduled visit during the screening phase;
   * Evidence of ventricular pre-excitation (e.g., Wolff Parkinson White syndrome);
   * Electrocardiographic evidence of either:

     * Complete left bundle branch block or right bundle branch block; OR
     * Incomplete left bundle branch block or right bundle branch block and QRS complex duration greater or equal to 120 msec on at least one ECG;
   * Having a pacemaker implant;
   * Congestive heart failure;
   * Evidence of second or third degree heart block;
   * Bradycardia as defined by sinus rate less than 50 bpm;
   * Personal or family history of Long QT Syndrome;
   * Personal history of arrhythmic cardiac disease, with the exception of sinus arrhythmia;
   * Personal history of syncope (i.e. cardiac syncope not including syncope due to vasovagal or epileptic causes).
8. Concurrent participation in another trial of any medication used or being studied for TB treatment, as defined in cited documents.
9. Is taking any medication that is contraindicated with the medicines in the trial regimen which cannot be stopped (with or without replacement) or requires a wash-out period longer than 2 weeks.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 754 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Week 73 Efficacy | Week 73 after randomization
  Proportion of participants with favorable outcome at week 73. A participant's outcome will be classified as favorable at week 73 if the outcome is not classified as unfavorable, and one of the following is true:
  * The last two culture results are negative. These two cultures must be taken from sputum samples collected on separate visits, the latest between weeks 65 and 73;
  * The last culture result (from a sputum sample collected between weeks 65 and 73) is negative; and either there is no other post-baseline culture result or the penultimate culture result is positive due to laboratory cross contamination; and bacteriological, radiological and clinical evolution is favorable;
  * There is no culture result from a sputum sample collected between weeks 65 and 73 or the result of that culture is positive due to laboratory cross contamination; and the most recent culture result is negative; and bacteriological, radiological and clinical evolution is favorable.

SECONDARY OUTCOMES:
Week 104 Efficacy | Week 104 after randomization
  Proportion of participants with favorable outcome at week 104.
  • A participant's outcome will be classified as favorable at week 104 if the outcome is not classified as unfavorable, and one of the following is true:
  1. The last two cultures are negative. These two cultures must be from sputum samples collected on separate visits, the latest between weeks 97 and 104;
  2. The last culture result (from a sputum sample collected between weeks 97 and 104) is negative; and either there is no other post-baseline culture result or the penultimate culture result is positive due to laboratory cross contamination; and bacteriological, radiological and clinical evolution is favorable;
  3. There is no culture result from a sputum sample collected between weeks 97 and 104 or the result of that culture is positive due to laboratory cross contamination; and the most recent culture result is negative; and bacteriological, radiological and clinical evolution is favorable.
Early Treatment Response (culture conversion) | Week 8 after randomization
  1. Proportion of patients with culture conversion assessed in MGIT system (and LJ where possible): 2 consecutive negative cultures from specimens collected at 2 different visits; if there is a missing or contaminated culture between 2 negatives, the definition of conversion is still met;
  2. Time to culture conversion: assessed in MGIT system (and LJ where possible): time from treatment initiation to first of 2 consecutive negative cultures; if there is a missing or contaminated culture between 2 negatives, the definition of conversion is still met;
  3. Change in time to positivity (TTP) in MGIT over 8 weeks.
Week 39 Efficacy | Week 39 after randomization
  Proportion of participants with favorable outcome at week 39:
  • A participant's outcome will be classified as favorable at week 39 if the last culture result (from a sample collected between weeks 36 and 39) is negative; and the outcome is not classified as unfavorable.
  A participant's outcome will be classified as unfavorable at week 39 in case of:
  1. In the experimental arm, addition or replacement of one or more drugs;
  2. In the control arm, addition or replacement of two or more drugs;
  3. Death from any cause;
  4. At least one culture result (from a sample collected between weeks 36 and 39) is positive;
  5. The patient is not assessable because the last available culture result is from a sample collected before week 36.
Week 73 Survival | Week 73 after randomization
  At 73 weeks, the proportion of patients who died of any cause
Week 104 Survival | Week 104 after randomization
  At 104 weeks, the proportion of patients who died of any cause
Week 73 Safety | Week 73 after randomization
  The proportion of participants with grade 3 or greater AEs and serious adverse events (SAEs) of any grade by 73 weeks
Week 104 Safety | Week 104 after randomization
  The proportion of participants with grade 3 or greater AEs and serious adverse events (SAEs) of any grade by 104 weeks
Week 73 Safety: proportion of patients with AESIs | Week 73 after randomization
  The proportion of patients with AESIs by 73 weeks
Week 104 Safety: proportion of patients with AESIs | Week 104 after randomization
  The proportion of patients with AESIs by 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Guglielmetti, MD, Principal Investigator — Médecins Sans Frontières, France; Carole Mitnick, Sc.D, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (12):
- National Center for Tuberculosis and Lung Diseases, Tbilisi, Georgia
- Aundh Chest Hospital, Pune, India
- Kazakhstan (3):
  - City Centre of Phthisiopulmonology, Almaty
  - Center of Phthisiopulmonology of Almaty Health Department, Almaty
  - National Center for Tuberculosis Problems, Almaty
- Partners In Health Lesostho, Maseru, Lesotho
- Pakistan (2):
  - The Indus Hospital, Karachi
  - Institute of Chest Disease,, Kotri
- Peru (3):
  - Centro de Investigación del Hospital Nacional Hipólito Unanue, Lima
  - Centro de Investigación de Enfermedades Neumológicas del Hospital Nacional Sergio Bernales, Lima
  - Hospital Nacional Dos de Mayo Parque Historia de la Medicina, Lima
- Medecins Sans Frontieres Belgium, Khayelitsha, South Africa

IPD SHARING:
Plan to Share IPD: Yes
After deidentification process most part of variables recorded in the eCRF (no patients name or ID, no site or country location, no dates but intervals from randomization, no birth dates but age at randomization, no information on staff...)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From Q4 2024 and will last 5 years renewable.
Access Criteria: * proposal has scientific value / the scientific question addresses a knowledge gap and avoids duplication without added value and unnecessary competition, and benefits the wider public health community
  * the data requested must be capable of answering the research question, and each variable requested must be required for the successful completion of the research
  * the methodology proposed to answer the research question must be sound
  * conform to the Data Access Guidelines, Ethics Framework, and Conflict of Interest Policy (see on website https://endtb.org/data-sharing-initiative)
URL: https://endtb.org/data-sharing-initiative

REFERENCES:
- [Derived] Guglielmetti L, Khan U, Velasquez GE, Gouillou M, Abubakirov A, Baudin E, Berikova E, Berry C, Bonnet M, Cellamare M, Chavan V, Cox V, Dakenova Z, de Jong BC, Ferlazzo G, Karabayev A, Kirakosyan O, Kiria N, Kunda M, Lachenal N, Lecca L, McIlleron H, Motta I, Toscano SM, Mushtaque H, Nahid P, Oyewusi L, Panda S, Patil S, Phillips PPJ, Ruiz J, Salahuddin N, Garavito ES, Seung KJ, Ticona E, Trippa L, Vasquez DEV, Wasserman S, Rich ML, Varaine F, Mitnick CD; endTB Clinical Trial Team. Oral Regimens for Rifampin-Resistant, Fluoroquinolone-Susceptible Tuberculosis. N Engl J Med. 2025 Jan 30;392(5):468-482. doi: 10.1056/NEJMoa2400327. PMID 39879593
- [Derived] Hewison C, Khan U, Bastard M, Lachenal N, Coutisson S, Osso E, Ahmed S, Khan P, Franke MF, Rich ML, Varaine F, Melikyan N, Seung KJ, Adenov M, Adnan S, Danielyan N, Islam S, Janmohamed A, Karakozian H, Kamene Kimenye M, Kirakosyan O, Kholikulov B, Krisnanda A, Kumsa A, Leblanc G, Lecca L, Nkuebe M, Mamsa S, Padayachee S, Thit P, Mitnick CD, Huerga H. Safety of Treatment Regimens Containing Bedaquiline and Delamanid in the endTB Cohort. Clin Infect Dis. 2022 Sep 29;75(6):1006-1013. doi: 10.1093/cid/ciac019. PMID 35028659
- [Derived] Guglielmetti L, Ardizzoni E, Atger M, Baudin E, Berikova E, Bonnet M, Chang E, Cloez S, Coit JM, Cox V, de Jong BC, Delifer C, Do JM, Tozzi DDS, Ducher V, Ferlazzo G, Gouillou M, Khan A, Khan U, Lachenal N, LaHood AN, Lecca L, Mazmanian M, McIlleron H, Moschioni M, O'Brien K, Okunbor O, Oyewusi L, Panda S, Patil SB, Phillips PPJ, Pichon L, Rupasinghe P, Rich ML, Saluhuddin N, Seung KJ, Tamirat M, Trippa L, Cellamare M, Velasquez GE, Wasserman S, Zimetbaum PJ, Varaine F, Mitnick CD. Evaluating newly approved drugs for multidrug-resistant tuberculosis (endTB): study protocol for an adaptive, multi-country randomized controlled trial. Trials. 2021 Sep 25;22(1):651. doi: 10.1186/s13063-021-05491-3. PMID 34563240
- [Derived] Seung KJ, Khan P, Franke MF, Ahmed S, Aiylchiev S, Alam M, Putri FA, Bastard M, Docteur W, Gottlieb G, Hewison C, Islam S, Khachatryan N, Kotrikadze T, Khan U, Kumsa A, Lecca L, Tassew YM, Melikyan N, Naing YY, Oyewusi L, Rich M, Wanjala S, Yedilbayev A, Huerga H, Mitnick CD. Culture Conversion at 6 Months in Patients Receiving Delamanid-containing Regimens for the Treatment of Multidrug-resistant Tuberculosis. Clin Infect Dis. 2020 Jul 11;71(2):415-418. doi: 10.1093/cid/ciz1084. PMID 31676905

DOCUMENTS (1):
  • Informed Consent Form (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT02754765/ICF_008.pdf